CLINICAL TRIAL: NCT07193511
Title: A Phase 1/2, First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of AVZO-103, a Nectin4/Trop2 ADC, as a Single Agent and in Combination Therapy in Patients With Locally Advanced or Metastatic Urothelial Cancer or Other Solid Tumors
Brief Title: Study of AVZO-103 as a Single Agent and in Combination Therapy in Patients With Locally Advanced or Metastatic Urothelial Cancer or Other Solid Tumors
Acronym: AVZO-103-1001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avenzo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVZO-103-1001
Record Dates: First submitted 2025-09-24; First posted 2025-09-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor Cancer; Locally Advanced; Metastatic Solid Tumors; Urothelial Cancer
Keywords: Solid Tumors; Metastatic; Locally Advanced; Urothelial Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1, monotherapy (Experimental): Part A
  Interventions: Drug: AVZO-103
- Phase 1, combination (Experimental): Part B
  Interventions: Drug: AVZO-103; Drug: Combination Agent
- Phase 2, monotherapy (Experimental): Part A
  Interventions: Drug: AVZO-103
- Phase 2, combination (Experimental): Part B
  Interventions: Drug: AVZO-103; Drug: Combination Agent

INTERVENTIONS:
Drug: AVZO-103 — Specific dose in protocol specified schedule
Drug: Combination Agent — Per label based on combination agent used
  Arms: Phase 1, combination; Phase 2, combination

SUMMARY:
This study, the first clinical trial of AVZO-103, aims to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, maximum tolerated dose, and antitumor activity of AVZO-103 when administered intravenously as a monotherapy and in combination therapy to patients with locally advanced or metastatic urothelial cancer or other solid tumors.

DETAILED DESCRIPTION:
Phase 1 is a dose escalation phase which will assess the safety and tolerability of AVZO-103 and determine the maximum tolerated dose (MTD) and preliminary recommended Phase 2 dose (RP2D) of AVZO-103 as a monotherapy. This data can guide selection of combination schedules and agents.

Phase 2 is a dose expansion phase that will aim to assess the antitumor activity of AVZO-103 as a monotherapy and in combination therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient must be an adult, 18 years of age and older with an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1 and a life expectancy of > 3 months.
* Patients with histologically or cytologically confirmed locally advanced/metastatic malignancies for tumor types of preferred indications:

  o Locally advanced or metastatic urothelial cancer and other solid tumors (as specified in the protocol).
* Measurable disease as assessed by Investigator using RECIST v1.1.
* Agree to provide molecular test report results to confirm eligibility and archival tumor samples and/or fresh biopsy, as applicable.
* Other protocol-defined Inclusion criteria apply.

Key Exclusion Criteria:

* Patients with active central nervous system (CNS) metastases are not eligible. Patients with asymptomatic and treated brain metastases may participate if they are radiologically stable for at least 4 weeks prior to the first dose of this study and do not require steroid treatment. Patients with suspected or confirmed leptomeningeal disease are not eligible, even if treated.
* Prior Stevens-Johnson syndrome/toxic epidermal necrolysis.
* History of drug-induced interstitial lung disease (ILD).
* History of any serious cardiovascular condition.
* Infection requiring IV antibiotics, antivirals, or antifungals within 2 weeks prior to first dose.
* History of allogenic stem cell or solid organ transplant.
* Other protocol-defined Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLTs) during the first cycle (Phase 1) | Approximately 2 years
  Number of participants with DLTs assessed for severity using CTCAE v5.0 criteria will be summarized by dose level.
Determine the maximum tolerated dose (MTD) and/or preliminary recommended Phase 2 dose (RP2D) (Phase 1) | Approximately 16 months
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and lab abnormalities (Phase 1) | From baseline until end of study treatment or study completion (approximately 2 years)
Objective Response Rate (ORR) (Phase 2) | From baseline through disease progression or study completion (approximately 2 years)
  Defined as the proportion of patients with a confirmed Complete Response (CR) or Partial Response (PR), as determined by the investigator by radiographic disease assessment according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Phase 1) | From baseline through disease progression or study completion (approximately 2 years)
Duration of Response (DOR) (Phase 1 and 2) | From baseline through disease progression or study completion (approximately 2 years)
  Defined as the time from the first confirmed response to radiologic/objective progression.
Disease Control Rate (DCR) (Phase 1 and 2) | From baseline through disease progression or study completion (approximately 2 years)
  Defined as the proportion of patients who achieve tumor response (CR or PR) and stable disease (SD) after treatment; calculated as the sum of CR, PR, and SD.
Progression Free Survival (PFS) (Phase 1 and 2) | From baseline through time to event on study or study completion (approximately 2 years)
  Defined as the time from study drug treatment to death or disease progression, as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Overall Survival (OS) (Phase 1 and 2) | Approximately 76 months
  Defined as the time from study drug treatment initiation to death from any cause.
PK Parameters: Maximum observed concentration (Cmax) (Phase 1) | Up to 2 years
PK Parameters: Minimum observed concentration (Cmin) (Phase 1) | Up to 2 years
PK Parameters: Time to maximum observed concentration (Tmax) (Phase 1) | Up to 2 years
PK Parameters: Elimination half-life (T1/2) (Phase 1) | Up to 2 years
PK Parameters: Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-last) (Phase 1) | Up to 2 years
PK Parameters: Area under the concentration-time curve from time 0 to infinity (AUCinf) (Phase 1) | Up to 2 years
PK Parameters: Area under the concentration-time curve from time 0 to the end of the dosing period (AUCτ) (Phase 1) | Up to 2 years
PK Parameters: Apparent Clearance (CL/F) (Phase 1) | Up to 2 years
PK Parameters: Apparent volume of distribution at steady-state (Vss) (Phase 1) | Up to 2 years
PK Parameters: Accumulation ratio (AR) (Phase 1) | Up to 2 years
Determination of RP2D (Phase 2) | Approximately 16 months
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and lab abnormalities (Phase 2) | From baseline until end of study treatment or study completion (approximately 2 years)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Avenzo Therapeutics Recruiting Site, Orlando, Florida
  - Avenzo Therapeutics Recruiting Site, Boston, Massachusetts
  - Avenzo Therapeutics Recruiting Site, Myrtle Beach, South Carolina
  - Avenzo Therapeutics Recruiting Site, Nashville, Tennessee
  - Avenzo Therapeutics Recruiting Site, Austin, Texas
  - Avenzo Therapeutics Recruiting Site, Irving, Texas